CLINICAL TRIAL: NCT03456648
Title: Apixaban in End-stage Kidney Disease : A Pharmacokinetics Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S57150; 2015-003132-12 (EudraCT Number); CV562247 (Other Grant/Funding Number: BMS)
Record Dates: First submitted 2017-02-20; First posted 2018-03-07 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-03

CONDITIONS: ESRD; Anticoagulant Toxicity
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: Single dose pharmacokinetics study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A : postdialysis low dose (Experimental): Interdialytic kinetics of low dose (2.5 mg apixaban) post-dialysis
  Interventions: Drug: apixaban
- Part A: ipostdialysis high dose (Experimental): Interdialytic kinetics of high dose (5 mg apixaban) post-dialysis
  Interventions: Drug: apixaban
- Part B : predialysis low dose (Experimental): Intra- and interrdialytic kinetics of low (2.5 mg) apixaban pre-dialysis
  Interventions: Drug: apixaban
- Part B : predialysis high dose (Experimental): Intra- and interrdialytic kinetics of high (5 mg) apixaban pre-dialysis
  Interventions: Drug: apixaban

INTERVENTIONS:
Drug: apixaban — non-vitamin K oral anticoagulant (NOAC)
  Other Names: Eliquis

SUMMARY:
Apixaban is a novel oral direct factor Xa inhibitor; In patients with atrial fibrillation, apixaban was superior to warfarin in preventing stroke or systemic embolism, caused less bleeding, and resulted in lower mortality (the ARISTOTLE trial). Given its favorable outcome profile compared to oral vitamin K antagonists in patients with normal kidney function and in patients with mild to moderate kidney disease and given the potential serious side-effects of oral vitamin K antagonists in end-stage kidney disease, apixaban may be an attractive alternative for systemic anticoagulation in dialysis patients. The pharmacokinetics of apixaban in end-stage renal disease is not well characterized.

The aim of the current study is to perform single dose pharmacokinetics / pharmacodynamics studies in patients treated with end-stage renal disease. The primary aim is to determine inter-dialytic pharmacokinetics of Apixaban, secondary aims are intra-dialytic pharmacokinetics and dose finding. Two doses of drugs will be studies (2.5 mg and 5 mg). Study drug will be administered at the end of a dialysis session (part A) and at the beginning of a dialysis session (Part B). Six (n=6) patients are scheduled to be included for each part and each dose.

Anti-Xa activity values (IIU/mL) will be converted to apixaban concentration data (ng/mL). Apixaban concentration-time profiles will be generated and observed values for the descriptive PK parameters Cmax (peak plasma concentration) and time to Cmax (Tmax) will be determined directly from these profiles. PK profiles will be further analyzed with non-compartmental analysis (NCA).

DETAILED DESCRIPTION:
RATIONALE

Chronic Kidney Disease (CKD) is one of the epidemics of modern times. In the recent National Health and Nutrition Examination Survey (NHANES), the overall prevalence of CKD (stages 1 to 4) increased from 10.0% in 1988-1994 to 13.1% in 1999-2004 (1). Mounting data point to the lethal synergy between chronic kidney disease (CKD) and cardiovascular disease (CVD) (2,3,4) Atrial fibrillation (AF) is an important co-morbid condition in patients with CKD. While prevalence differs from region to region, it is estimated that between 5 and 10% of dialysis patients have AF (5). Analyses of the US renal data system (USRDS) demonstrate that the prevalence of AF in patients with hemodialysis continues to rise (6). Prevalent AF is positively associated with all-cause mortality and stroke, similar to that of the general population (5).

The choice of the optimal anticoagulation regimen for hemodialysis patients with AF is hampered by lack of randomized controlled trials. Observational data support the use of the CHADS2-score for risk stratification of AF in HD (5). Cost-utility analyses suggest that warfarin appears to be the optimal therapy to prevent thromboembolic stroke in hemodialysis patients with AF (7). These analyses however extrapolate the decrease in risk of stroke observed in randomized trials of oral vitamin K antagonist therapy in the general population (7). Both retrospective and prospective observational data however observe an increased risk for stroke in HD patients receiving oral vitamin K antagonist therapy for AF (8,5).

Recent findings shed a worrisome light on the pleiotropic effects of oral vitamin K antagonist therapy in patients with advanced chronic kidney disease. Besides promoting undercarboxylation of the pro- and anticoagulant factors (II, VII, IX, X, protein S, protein C) several other glutamine-domain containing proteins remain undercarboxylated. Matrix-Gla protein is a powerful calcification inhibitor. Nonphosphorylated matrix-Gla protein has been associated with overall mortality and cardiovascular mortality in HD patients (9). Observational data suggest that patients treated with oral vitamin K antagonists demonstrate higher valvular and coronary calcium (10). Prospective trials currently investigate the effects of vitamin K supplementation on the evolution of vascular calcification in patients with end-stage kidney disease and on aortic valve calcifications.

Apixaban is a novel oral direct factor Xa inhibitor; In patients with atrial fibrillation, apixaban was superior to warfarin in preventing stroke or systemic embolism, caused less bleeding, and resulted in lower mortality (the ARISTOTLE trial) (11). An important benefit of apixaban as compared to other recent NOACs, e.g. dabigatran and rivaroxaban, is that the elimination is less dependent on kidney function as only 25% is excreted renally and 75% is excreted through the hepatobiliary system, with a mean elimination half-life of 8-15 hours in healthy adults.

Given its favorable outcome profile compared to oral vitamin K antagonists in patients with normal kidney function and in patients with mild to moderate kidney disease and given the potential serious side-effects of oral vitamin K antagonists in end-stage kidney disease, apixaban may be an attractive alternative for systemic anticoagulation in dialysis patients. The pharmacokinetics of apixaban in end-stage renal disease is not well characterized.

HYPOTHESIS The pharmacokinetics profile of apixaban allows safe use in patients with end-stage renal disease

STUDY DESIGN Open label non-randomized phase II pharmacokinetics study.

STUDY AIMS

Primary:

To determine inter-dialytic pharmacokinetics of Apixaban

Secondary:

* To determine intra-dialytic pharmacokinetics of Apixaban
* Dose finding of apixaban in patients treated with hemodialysis

DOSING AND TIMING Part A - interdialytic kinetics Dose titration

1. single dose 2.5 mg post-dialysis
2. single dose 5 mg post-dialysis As study drug is administered immediately following dialysis, part A will provide inter-dialytic PK data (primary aim)

Part B - intra- plus interdialytic pharmacokinetics Dose titration

1. single dose 2.5 mg 30 minutes pre-dialysis
2. single dose 5 mg 30 minutes pre-dialysis As study drug is administered 30 minutes pre-dialysis, part B will provide intra-dialytic kinetic PK data (secondary aim). As we expect that study drug effect is not completely lost at the end of the dialysis session, we will continue sampling blood at fixed time-points after end of dialysis. These data may contribute to interdialytic PK (primary study aim).

NUMBER OF STUDY PARTICIPANTS

We aim to include 6 patients for each part and dosage:

Part A - Interdialytic kinetics 2.5 mg N = 6 5 mg N = 6

Part B - Intra- plus interdialytic kinetics 2.5 mg N = 6 5 mg N = 6

Based on previous publications on single dose pharmacokinetics of apixaban in healthy volunteers (12), we expect that 6 patients per part will provide sufficient data to generate PK profiles.

SCHEDULED BLOOD SAMPLING

Part A - Interdialytic kinetics (post-dialysis dosing)

* Sampling at start of first dialysis (pre)
* Sampling at end of dialysis (post, t = 0)
* Sampling for pharmacokinetics (t =0.5, 1, 2, 4, 8, 24 hours post dialysis)
* Sampling at start of second dialysis (t = 44 hours)
* Sampling at end of second dialysis (t = 48 hours)

Part B - Intradialytic kinetics (pre-dialysis dosing)

* Sampling at start of first dialysis (pre)
* Sampling for pharmacokinetics ( t=0.25, 0.5, 1, 1.5,2, 3,4 hours after dialysis start)
* Sampling at end of dialysis (post, t = 0)
* Sampling for pharmacokinetics (t =0.5, 1, 2, 4, 24 hours post dialysis)
* Sampling at start of second dialysis (t = 44 hours)
* Sampling at end of second dialysis (t = 48 hours)

ANALYTICAL TECHNIQUES

Apixaban concentrations (ng/mL) will be determined based on a calibration curve with Apixaban (Apixaban Calibrator and controls, Hyphen).

Conventional anticoagulation used for hemodialysis is by heparin or low molecular weight heparins (LMWH). This will lead to significant interference with the proposed chromogenic anti-Xa activity assays. To exclude interference of anticoagulation for hemodialysis during the study period, the routine anticoagulation will be switched to regional citrate anticoagulation according to local protocol during the study period. The following will be applied.

* One week wash-out period of (low molecular weight) heparin, during which hemodialysis anticoagulation is according to the local regional citrate anticoagulation protocol (no use of (low molecular weight) heparins).
* During the study period hemodialysis anticoagulation is according to the local regional citrate anticoagulation protocol (no use of (low molecular weight) heparins).

PHARMACOKINETICS ANALYSES

Anti-Xa activity values (IIU/mL) will be converted to apixaban concentration data (ng/mL) based on the previously demonstrated linear relationship (e.g. Frost et al., 2014 - PMID: 24697979). Apixaban concentration-time profiles will be generated and observed values for the descriptive PK parameters Cmax (peak plasma concentration) and time to Cmax (Tmax) will be determined directly from these profiles. PK profiles will be further analyzed with non-compartmental analysis (NCA). Briefly, the slope (λ) of the terminal phase of the concentration-time profile will be determined by log-linear regression on the appropriate number (typically at least 3) of data points. The terminal (elimination) half-life (t1/2, λ) will be calculated from Ln(2)/λ. The area under the curve (AUC) between administration (time 0) and the last measurable data point (AUC0-T) will be calculated with the 'Lin up/Log down' trapezoidal method. The AUCT-∞ will be obtained from the last measureable concentration divided by λ, and will be summed with AUC0-T to obtain AUC0-∞ (total exposure). Similarly, after plotting plasma concentration-time products as a function of time, Area under the first Moment Curve (AUMC) values will be calculated. The mean residence time (MRT, h) will be obtained from AUMC/AUC. Mean half-life (t1/2) will be calculated as Ln(2)×MRT. Oral ('apparent') clearance (Cl/F) values will be obtained by dividing dose by AUC. The volume of distribution at steady (Vdss/F) will be obtained as MRT x Cl/F. As alternative to NCA, the feasibility of analyzing the data with a 1-compartmental model with first order absorption will be explored as well. Summary statistics will be tabulated for all relevant PK parameters: (i) the descriptive parameters Cmax, Tmax and AUC0-∞ (total exposure), (ii) MRT and mean t1/2, (iii) the primary (fundamental) PK parameters Cl/F and Vd/F. Reported parameters will enable appropriate comparison with previously published data on apixaban PK in various populations. For the purpose of dose finding, AUC0-∞ (total exposure) represents the key parameter.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 85 years
* Treated with maintenance (dialysis vintage >3 months) thrice weekly hemodialysis
* Written and signed informed consent

Exclusion Criteria:

* Treated with oral vitamin K antagonists
* Recent (< 4 weeks prior to informed consent) major surgery
* Recent (< 4 weeks prior to informed consent) severe bleeding episode requiring blood transfusion and/ or hospitalization
* Concurrent moderate to severe liver dysfunction
* Participation in an interventional study with investigational medication

For women of childbearing potential the following criteria apply:

* A women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes. In addition, females under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40mIU/mL to confirm menopause.
* Females treated with hormone replacement therapy, (HRT) are likely to have artificially suppressed FSH levels and may require a washout period in order to obtain a physiologic FSH level. The duration of the washout period is a function of the type of HRT used. The duration of the washout period below are suggested guidelines and the investigators should use their judgement in checking serum FSH levels. If the serum FSH level is >40 mIU/ml at any time during the washout period, the woman can be considered postmenopausal :

  * 1 week minimum for vaginal hormonal products (rings, creams, gels)
  * 4 week minimum for transdermal products
  * 8 week minimum for oral products Other parenteral products may require washout periods as long as 6 months.

    1. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study drug.
    2. Women must not be breastfeeding
    3. WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug Apixaban plus 5 half-lives of study drug (3 days) plus 30 days (duration of ovulatory cycle) for a total of 33 days post-treatment completion.
    4. Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug Apixaban plus 5 half-lives of the study drug (3 days) plus 90 days (duration of sperm turnover) for a total of 93 days post-treatment completion.
    5. Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However they must still undergo pregnancy testing as described in this section.

Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly. At a minimum, subjects must agree to the use of one method of highly effective contraception as listed below:

* Male condoms with spermicide
* Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) such as Mirena by WOCBP subject or male subject's WOCBP partner. Female partners of male subjects participating in the study may use hormone based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug
* IUDs, such as ParaGard
* Tubal ligation
* Vasectomy.
* Complete Abstinence Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Female subjects must continue to have pregnancy tests. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-25 (Actual); Primary Completion 2018-08-24 (Actual); Study Completion 2018-08-24 (Actual)

PRIMARY OUTCOMES:
AUC0-T apixaban | 48 hours
  Anti-Xa activity values (IIU/mL) will be converted to apixaban concentration data (ng/mL) based on the previously demonstrated linear relationship (e.g. Frost et al., 2014 - PMID: 24697979).
  The area under the curve (AUC) between administration (time 0) and the last measurable data point (AUC0-T) will be calculated with the 'Lin up/Log down' trapezoidal method. The AUCT-∞ will be obtained from the last measureable concentration divided by λ, and will be summed with AUC0-T to obtain AUC0-∞ (total exposure).
  the slope (λ) of the terminal phase of the concentration-time profile will be determined by log-linear regression on the appropriate number (typically at least 3) of data points. The terminal (elimination) half-life (t1/2, λ) will be calculated from Ln(2)/λ.
Cmax | 48 hours
  Apixaban concentration-time profiles will be generated and observed values for the descriptive PK parameter Cmax (peak plasma concentration) will be determined directly from the time-concentration curve
Tmax | 48 hours
  Apixaban concentration-time profiles will be generated and observed values for the descriptive PK parameter time to Cmax (Tmax)) will be determined directly from the time-concentration curve

SECONDARY OUTCOMES:
Occurrence of SAE | 48 hours
  Occurrence of serious adverse events (SAE) will be analyzed as an important safety variable

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Vlaams-brabant, Belgium

IPD SHARING:
Plan to Share IPD: No